CLINICAL TRIAL: NCT04575935
Title: Laparoscopic Cytoreduction After Neoadjuvant Chemotherapy
Brief Title: Minimally Invasive Surgery After Neoadjuvant Chemotherapy for the Treatment of Stage IIIC-IV Ovarian, Primary Peritoneal, or Fallopian Tube Cancer, LANCE Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-0165; NCI-2020-04165 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0165 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-09-08; First posted 2020-10-05 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Advanced Ovarian Carcinoma; Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Tumor; Fallopian Tube Serous Neoplasm; Fallopian Tube Transitional Cell Carcinoma; Ovarian Clear Cell Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Serous Adenocarcinoma; Ovarian Transitional Cell Carcinoma; Primary Peritoneal Clear Cell Adenocarcinoma; Primary Peritoneal Endometrioid Adenocarcinoma; Primary Peritoneal Serous Adenocarcinoma; Primary Peritoneal Transitional Cell Carcinoma; Stage IIIC Fallopian Tube Cancer AJCC v8; Stage IIIC Ovarian Cancer AJCC v8; Stage IIIC Primary Peritoneal Cancer AJCC v8; Stage IV Fallopian Tube Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Primary Peritoneal Cancer AJCC v8; Stage IVA Fallopian Tube Cancer AJCC v8; Stage IVA Ovarian Cancer AJCC v8; Stage IVA Primary Peritoneal Cancer AJCC v8; Stage IVB Fallopian Tube Cancer AJCC v8; Stage IVB Ovarian Cancer AJCC v8; Stage IVB Primary Peritoneal Cancer AJCC v8
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Drug Therapy; Laparotomy; Minimally Invasive Surgical Procedures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (MIS, standard of care chemotherapy) (Experimental): Patients undergo MIS within 6 weeks after last cycle of standard of care neoadjuvant chemotherapy. If during MIS the surgeon thinks complete gross resection can only be accomplished by performing an open procedure, patients may undergo laparotomy instead. Within 6 weeks after surgery, patients receive standard of care chemotherapy.
  Interventions: Drug: Chemotherapy; Procedure: Minimally Invasive Surgery; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm B (laparotomy, standard of care chemotherapy) (Active Comparator): Patients undergo laparotomy within 6 weeks after last cycle of standard of care neoadjuvant chemotherapy. Within 6 weeks after surgery, patients receive standard of care chemotherapy.
  Interventions: Drug: Chemotherapy; Procedure: Laparotomy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Chemotherapy — Receive standard of care chemotherapy
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
Procedure: Laparotomy — Undergo laparotomy
  Arms: Arm B (laparotomy, standard of care chemotherapy)
Procedure: Minimally Invasive Surgery — Undergo MIS
  Other Names: Minimally-Invasive Surgery
  Arms: Arm A (MIS, standard of care chemotherapy)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial compares minimally invasive surgery (MIS) to laparotomy in treating patients with stage IIIC-IV ovarian, primary peritoneal, or fallopian tube cancer who are receiving chemotherapy before and after surgery (neoadjuvant chemotherapy). MIS is a surgical procedure that uses small incision(s) and is intended to produce minimal blood loss and pain for the patient. Laparotomy is a surgical procedure which allows the doctors to remove some or all of the tumor and check if the disease has spread to other organs in the body. MIS may work the same or better than standard laparotomy after chemotherapy in prolonging the return of the disease and/or improving quality of life after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To examine whether MIS is non-inferior to laparotomy in terms of disease free survival (DFS) in women with advanced stage epithelial ovarian cancer (EOC) that received 3 to 4 cycles of neoadjuvant chemotherapy (NACT).

SECONDARY OBJECTIVES:

I. To determine if there are differences in health-related quality of life (HR-QoL) in patients undergoing MIS versus (vs) laparotomy as assessed with the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30), QLQ-Ovarian Cancer Module (OV28), and Functional Assessment of Cancer Therapy-General (FACT-G7).

II. To determine if there are differences between patients undergoing MIS vs laparotomy in the rate of optimal cytoreduction (defined as residual tumor nodules each measuring 1 cm or less in maximum diameter) and complete cytoreduction (defined as no evidence of macroscopic disease).

III. To examine whether MIS is non-inferior to laparotomy in terms of overall survival (OS) in women with advanced stage EOC that received 3 to 4 cycles of NACT.

IV. To determine if there are differences between patients undergoing MIS vs laparotomy in surgical morbidity and mortality, intraoperative injuries, and post-operative complications.

V. To determine the rates of MIS converted to laparotomy and the reasons.

VI. To determine if there are any difference in costs and cost-effectiveness between patients undergoing MIS vs laparotomy.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients undergo MIS within 6 weeks after last cycle of standard of care neoadjuvant chemotherapy. If during MIS the surgeon thinks complete gross resection can only be accomplished by performing an open procedure, patients may undergo laparotomy instead. Within 6 weeks after surgery, patients receive standard of care chemotherapy.

ARM B: Patients undergo laparotomy within 6 weeks after last cycle of standard of care neoadjuvant chemotherapy. Within 6 weeks after surgery, patients receive standard of care chemotherapy.

After completion of study, patients are followed up within 6 weeks of completing post-surgery chemotherapy, then every 3 months for the first 2 years, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Stage IIIC or IV, high-grade (serous, endometrioid, clear-cell, transitional carcinomas), invasive epithelial ovarian carcinoma, primary peritoneal carcinoma, or fallopian-tube carcinoma or pathology consistent with high-grade mullerian carcinoma.
* Patient is considered by treating physician to be a surgical candidate after completion of 3 to 4 cycles of platinum-based chemotherapy, or an investigational neoadjuvant regimen given according to protocol, with complete radiologic resolution of any disease outside the abdominal cavity. Pleural effusions are acceptable per the local PI's discretion.
* Normalization of CA-125 according to individual participating center reference range (Note: Among patients with a normal CA-125 at initiation of therapy, the CA-125 cannot exceed 35 U/mL at the completion of NACT prior to interval debulking surgery.) or has a CA-125 value ≤500 and is scheduled to undergo a diagnostic laparoscopy prior to debulking surgery. a. For patients undergoing diagnostic laparoscopy, surgeon considers that optimal debulking is feasible either by MIS or laparotomy.
* Timeframe of < 6 weeks (42 days) from the last cycle of NACT to interval debulking surgery. Overall timeframe may be extended per MD Anderson PI discretion.
* ECOG performance status 0-2
* Signed informed consent and ability to comply with follow-up
* Negative pregnancy test by blood or urine (within 14 days prior to surgery)
* Disease free of other active malignancies in the previous five years, except basal and squamous cell carcinomas of the skin

Exclusion Criteria:

* Evidence of tumor not amenable to minimally invasive resection on pre-operative imaging (CT, PET-CT, or MRI) including but not limited to the following findings that may preclude minimally invasive resection per surgeon's assessment. • Failure of improvement of ascites during NACT (trace ascites is allowed) • Small bowel or gastric tumor involvement • Colon or rectal tumor involvement • Diaphragmatic tumor involvement • Splenic or hepatic surface or parenchymal tumor involvement • Mesenteric tumor involvement • Tumor infiltration of the lesser peritoneal sac
* History of psychological, familial, sociological or geographical condition potentially preventing compliance with the study protocol and follow-up schedule
* Inability to tolerate prolonged Trendelenburg position or pneumoperitoneum as deemed by participating institution's clinicians
* Any other contraindication to MIS as assessed by the clinician

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2020-08-05 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | Between randomization and physical or radiographic evidence of recurrence (local/distant) or death (all causes), assessed up to 5 years
  Kaplan Meier curves will be used to describe DFS over time. Log-rank test will be used to compare DFS between the control and experimental arms. The treatment effects will be summarized by means of a hazard ratio with its associated 95% confidence interval. Two years DFS rate will be computed with a targeted 95% confidence interval (CI).

SECONDARY OUTCOMES:
Health related-quality of life (HR-QoL) | Up to 1 year post surgery chemotherapy
  HR-QoL of patients will be assessed with European Organization for Research and Treatment of Cancer (EORTC Scale 1-Not at all, 2-A little bit, 3-Quite a bit, 4-Very Much)
Health related-quality of life (HR-QoL) | Up to 1 year post surgery chemotherapy
  HR-QoL of patients will be assessed Quality of Life Questionnaire-Core 30 (QLQC30 scale 1-Not at all, 2-A little bit, 3-Quite a bit, 4-Very Much)
Health related-quality of life (HR-QoL) | Up to 1 year post surgery chemotherapy
  HR-QoL of patients will be assessed with QLQ-Ovarian Cancer Module (OV28 Scale 1- Not at all, 2- A little bit, 3-Quite a bit, 4-Very Much).) (ovarian supplement)
Health related-quality of life (HR-QoL) | Up to 1 year post surgery chemotherapy
  HR-QoL of patients will be assessed with Functional Assessment of Cancer Therapy-General short-form (FACT-G7 Scale 1- Not at all, 2- A little bit, 3-Quite a bit, 4-Very Much).
Optimal cytoreduction | At the end of surgery
  Defined as residual tumor nodules each measuring 1 cm or less in maximum diameter.
Complete cytoreduction | At the end of surgery
  Defined as no evidence of macroscopic disease.
Overall survival (OS) | Between randomization and death (all causes), assessed up to 5 years
  Overall survival will be estimated using the Kaplan-Meier method, and will be described using the median with its 95% CI. Univariate Cox proportional hazards model (i.e., logrank test) will be used to estimate hazard ratios (HR: control arm versus investigational arm) with a 95% CI. When appropriate, multivariate Cox analyses will be performed, in which a univariate selection procedure will serve to identify eligible explanatory variables with univariate Cox (using Wald test) p-value lower than 0.10 as potential prognostic value. Follow-up will be estimated using the reverse Kaplan-Meier method, and will be described using the median with its 95% CI.
Surgical morbidity | Up to 6 months post surgery
  Rates of surgical complications according to Surgical morbidity (Common Terminology Criteria for Adverse Events [CTCAE] version [v] 5.0 & Clavien Dindo classification and mortality (30-day post-operative for adverse events and up to 6 months post-operative for adverse events of interest).
Mortality | Up to 6 months post surgery
  Mortality rates (Common Terminology Criteria for Adverse Events [CTCAE] version [v] 5.0 & Clavien Dindo classification and mortality (30-day post-operative for adverse events and up to 6 months post-operative for adverse events of interest).
Intraoperative injuries | During surgery
  Coded as yes or no and categorized as involving the bowel, veins, arteries, ureter, bladder, or other site.
Minimally invasive surgery (MIS) converted to laparotomy | During surgery
  Prospectively completed forms documented reasons for conversion of MIS to laparotomy.
Cost of the procedure | Up to 6 months post surgery
  A cost analysis may be performed in some countries.

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Rauh-Hain, Principal Investigator — M.D. Anderson Cancer Center
Locations (19):
- United States (13):
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Cleveland Clinic Foundation - Florida, Weston, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - NYU Langone Health, Mineola, New York
  - Columbia University Medical Center, New York, New York
  - Duke, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Lyndon Baines Johnson General, Houston, Texas
  - Houston Methodist, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Canada (2):
  - Arthur J.E. Child Comprehensive Cancer Centre - Calgary, Calgary
  - University Health Network - Princess Margaret Cancer Centre, Toronto
- Italy (2):
  - Sant'Orsola Hospital di Bologna, Bologna
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
- Instituto Nacional de Cancerología (Mexico), Tlalpan, Mexico
- Amsterdam UMC - Locatie AMC | H5Zuid 154, Amsterdam, Netherlands

REFERENCES:
- [Derived] Rauh-Hain JA, Melamed A, Pareja R, May T, Sinno A, McNally L, Horowitz NS, De Iaco P, Michener CM, Van Lonkhuijzen L, Iniesta MD, Yuan Y, Ramirez PT, Fagotti A. Laparoscopic Cytoreduction After Neoadjuvant Chemotherapy in High-Grade Epithelial Ovarian Cancer: A LANCE Randomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2446325. doi: 10.1001/jamanetworkopen.2024.46325. PMID 39570589
- See also: MD Anderson Cancer Center — http://www.mdanderson.org